CLINICAL TRIAL: NCT00569491
Title: TAXUS ARRIVE: TAXUS Peri-Approval Registry: A Multi-Center Safety Surveillance Program
Acronym: ARRIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Kellie Windle, Clinical Project Manager, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2021
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: TAXUS Express 2™ — TAXUS Express™ Paclitaxel-Eluting Coronary Stent System

SUMMARY:
The TAXUS ARRIVE study is a multi-center safety and surveillance study designed to to compile safety surveillance and clinical outcomes data for the TAXUS™ Express2™ Paclitaxel-Eluting Coronary Stent System in routine clinical practice and to identify low frequency TAXUS related clinical events.

ELIGIBILITY:
Appropriate Patient Criteria:

* Patient is eligible to receive a Boston Scientific TAXUS Stent.

Inappropriate Patients Criteria:

* Known sensitivity to paclitaxel.
* Known allergy to stainless steel.
* Patients in whom antiplatelet and / or anticoagulant therapy is contraindicated.
* Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon or proper placement of the stent or delivery device.
* Patients with unresolved vessel thrombus at the lesion site.
* Patients with coronary artery reference vessel diameters < 2.5 mm or > 3.75 mm.
* Patients with lesions located in the left main coronary artery, ostial lesions, or lesions located at a bifurcation.
* Patients with diffuse disease or poor overflow distal to the identified lesions.
* Patients with tortuous vessels in the region of the obstruction or proximal to the lesion.
* Patients with a recent acute myocardial infarction where there is evidence of thrombus or poor flow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2585 (Actual)
Dates: Start 2004-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Rate of TAXUS stent related cardiac events at a 1-year post implant procedure as classified by the Clinical Events Committee | 1 year post-implant procedure

SECONDARY OUTCOMES:
Rate of TAXUS stent related cardiac events as classified by the Clinical Events Committee | 30 days, 6 months, 2 years post-implant procedure
Rate of target vessel related cardiac events as classified by the Clinical Events Committee | 30 days, 6 months, 1 and 2 years post-implant procedure
Rate of other TAXUS related events | 30 days, 6 months, 1 and 2 years post-implant procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Rose, MS, Study Director — Boston Scientific Corporation; John M Lasala, MD, PhD, Principal Investigator — Washington University School of Medicine; David A Cox, MD, Principal Investigator — Lehigh Valley Physician Group
Locations (50):
- United States (50):
  - Advanced Cardiac Specialists, Gilbert, Arizona
  - Cardiology Associates of NEA, Jonesboro, Arkansas
  - University of California Davis Medical Center, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Good Samaritan, San Jose, California
  - Little Company of Mary Hospital, Torrance, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Advanced Clinical Research Group, LLC, Juniper, Florida
  - Florida Heart Institute, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Georgia Heart and Vascular Center, Macon, Georgia
  - Alexian Brothers Medical Center, Elk Grove, Illinois
  - Lutheran Hospital/NIRA, Fort Wayne, Indiana
  - St Francis Hospital, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Our Lady of Lourdes, Lafayette, Louisiana
  - Willis Knighton Medical Center, Shreveport, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - Delmarva Heart Research Foundation, Inc, Salisbury, Maryland
  - Regional Cardiology Associates, Grand Blanc, Michigan
  - Metro Cardiology Consultants, Coon Rapids, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cardiovascular Consultants of Nevada, Las Vegas, Nevada
  - Morristown Memorial, Morristown, New Jersey
  - Westchester County Medical Center, Valhalla, New York
  - Asheville Cardiology Associates, PA, Asheville, North Carolina
  - Mid-Carolina Cardiology Presbyterian Hospital, Charlotte, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - WakeMed - Wake Heart Associates, Raleigh, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Cleveland Cardiovascular Research Foundation, Fairview Park, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Presbyterian University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Greenville Hospital Systems, Greenville, South Carolina
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Cardiovascular Associates, PC, Kingsport, Tennessee
  - Methodist Dallas Medical Center, Dallas, Texas
  - Texas Cardiac Center, Lubbock, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Trinity Mother Frances Hospital, Tyler, Texas
  - Clear Lake Regional Medical Center, Webster, Texas
  - LDS Hospital, Salt Lake City, Utah
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Hope Heart Institute, Bellevue, Washington
  - St. Peters Hospital, Olympia, Washington
  - St Mary's Hospital, Huntington, West Virginia
  - Care Foundation, Inc., Wausau, Wisconsin

REFERENCES:
- [Derived] Brilakis ES, Lasala JM, Cox DA, Berger PB, Bowman TS, Starzyk RM, Dawkins KD. Outcomes after implantation of the TAXUS paclitaxel-eluting stent in saphenous vein graft lesions: results from the ARRIVE (TAXUS Peri-Approval Registry: A Multicenter Safety Surveillance) program. JACC Cardiovasc Interv. 2010 Jul;3(7):742-50. doi: 10.1016/j.jcin.2010.04.012. PMID 20650436
- [Derived] Lasala JM, Cox DA, Dobies D, Baran K, Bachinsky WB, Rogers EW, Breall JA, Lewis DH, Song A, Starzyk RM, Mascioli SR, Dawkins KD, Baim DS; ARRIVE 1 and ARRIVE 2 Participating Physicians. Drug-eluting stent thrombosis in routine clinical practice: two-year outcomes and predictors from the TAXUS ARRIVE registries. Circ Cardiovasc Interv. 2009 Aug;2(4):285-93. doi: 10.1161/CIRCINTERVENTIONS.109.852178.109.852178. Epub 2009 Jul 22. PMID 20031730
- [Derived] Lasala JM, Cox DA, Lewis SJ, Tadros PN, Haas RC, Schweiger MJ, Chhabra A, Untereker WJ, Starzyk RM, Mascioli SR, Dawkins KD, Baim DS. Expanded use of the TAXUS Express Stent: two-year safety insights from the 7,500 patient ARRIVE Registry programme. EuroIntervention. 2009 May;5(1):67-77. doi: 10.4244/eijv5i1a11. PMID 19577985